CLINICAL TRIAL: NCT02262780
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses (40 mg Telmisartan / 12.5 mg HCTZ to 80 mg Telmisartan / 12.5 mg HCTZ) and Multiple Oral Doses (80 mg Telmisartan / 12.5 mg HCTZ) of Drug in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising and Multiple Oral Doses of Telmisartan / Hydrochlorothiazide (HCTZ) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.453
Record Dates: First submitted 2014-10-10; First posted 2014-10-13 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Hydrochlorothiazide

ARMS (3):
- Single low dose Telmisartan with HCTZ (Experimental)
  Interventions: Drug: Low dose of telmisartan; Drug: HCTZ
- Single high dose Telmisartan with HCTZ (Experimental)
  Interventions: Drug: High dose of telmisartan; Drug: HCTZ
- Multiple high dose Telmisartan with HCTZ (Experimental)
  Interventions: Drug: High dose of telmisartan; Drug: HCTZ

INTERVENTIONS:
Drug: Low dose of telmisartan
  Arms: Single low dose Telmisartan with HCTZ
Drug: High dose of telmisartan
  Arms: Multiple high dose Telmisartan with HCTZ; Single high dose Telmisartan with HCTZ
Drug: HCTZ

SUMMARY:
Group 1:

To investigate safety, tolerability and pharmacokinetics of Telmisartan + HCTZ (T40/H12.5 and T80/H12.5)

Group 2:

To investigate safety, tolerability and pharmacokinetics of Telmisartan + HCTZ (T80/H12.5 x 7 days)

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: No finding deviating of clinical relevance and no evidence of a clinically relevant concomitant disease based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature), 12-lead ECG, clinical laboratory tests
* Age ≥20 and Age ≤35 years
* Body Mass Index (BMI) ≥17.6 and BMI ≤26.4 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with "Good Clinical Practice (GCP)"

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* Any laboratory value outside the reference range that is of clinical relevance
* Positive result for hepatitis B surface (HBs) antigen, anti hepatitis C virus (HCV) antibodies, Syphilitic test or HIV test
* Surgery of gastrointestinal tract (except appendectomy)
* History of relevant orthostatic hypotension (mean standing SBP varies by ≥ 20 mmHg from mean supine systolic blood pressure (SBP) and/or mean standing diastolic blood pressure (DBP) varies by ≥ 10 mmHg from mean supine DBP), fainting spells or blackouts.
* History of hepatic dysfunction (e.g. biliary cirrhosis, cholestasis)
* History of serious renal dysfunction
* History of bilateral renal artery stenosis or renal artery stenosis in a solitary kidney
* History of cerebrovascular disorder
* History of hyperkalemia
* Known hypersensitivity to any component of the formulation; known hypersensitivity to any other angiotensin II receptor antagonist; known hypersensitivity to sulfonamides or sulphonamide-derived drugs (e.g. thiazides)
* History of impaired glucose tolerance
* History of hypokalemia
* History of hyperuricemia
* Salt restriction therapy
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 7 days prior to administration or during the trial
* Participation in another trial with an investigational drug within four months or 6 half-lives of the investigational drug, whichever is longer, prior to administration or during the trial
* Smoker (more than 20 cigarettes /day)
* Alcohol abuse
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within seven days prior to administration)
* Intake of alcohol within two days prior to administration
* Inability to comply with dietary regimen of study centre
* Inability to comply with smoking cessation during hospitalization

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-12-01 (Actual); Primary Completion 2004-02-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically relevant findings in physical examination | up to 10 days after last drug administration
Number of patients with clinically relevant findings in vital signs | up to 10 days after last drug administration
  blood pressure, pulse rate, body temperature
Number of patients with clinically relevant findings in 12-lead ECG | up to 10 days after last drug administration
Number of patients with clinically relevant findings in clinical laboratory tests | up to 10 days after last drug administration
Number of patients with adverse events | up to 10 days after last drug administration
Global assessment of tolerability by the investigator | up to 10 days after last drug administration
  verbal rating scale

SECONDARY OUTCOMES:
Maximum concentration of the analytes in plasma (Cmax) | Up to 96 hours after drug administration
Area under the concentration time curve of the analytes in plasma (AUC) | Up to 96 hours after drug administration
Time from dosing to maximum concentration of the analytes in plasma (tmax) | Up to 96 hours after drug administration
Terminal rate constant of the analytes in plasma (λz) | Up to 96 hours after drug administration
Terminal half-life of the analytes in plasma (t1/2) | Up to 96 hours after drug administration
Mean residence time of the analytes in the body after po administration (MRTpo) | Up to 96 hours after drug administration
Apparent clearance of the analytes in the plasma after extravascular administration (CL/F) | Up to 96 hours after drug administration
Apparent volume of distribution of the analytes in plasma during the terminal phase λz following an extravascular dose (Vz/F) | Up to 96 hours after drug administration
Amount of HCTZ that is eliminated in urine from the time interval t1 to t2 (Aet1-t2) | Up to 48 hours after drug administration
Fraction of HCTZ excreted unchanged in urine from time point t1 to t2 (fet1-t2) | Up to 48 hours after drug administration
Renal clearance of HCTZ in plasma from the time point t1 until the time point t2 (CLR, t1-t2) | Up to 48 hours after drug administration
Minimum measured concentration of the analytes in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | Up to 96 hours after drug administration
Average concentration of the analytes in plasma at steady state (Cavg) | Up to 96 hours after drug administration
Accumulation ratio of the analytes in plasma after multiple dose administration over a uniform dosing interval τ (RA) | Up to 96 hours after drug administration